CLINICAL TRIAL: NCT00532233
Title: A Open-label, Multicenter Study, With a Single Intravenous Dose of QAX576 to Determine IL-13 Production in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: SD, IL-13 Production Rate in IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CQAX576A2202; NCT00843999 (obsolete NCT alias)
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): QAX576
  Interventions: Drug: QAX576

INTERVENTIONS:
Drug: QAX576

SUMMARY:
The purpose of this study is to investigate how QAX576 affects levels of interleukin 13 (IL-13) in patients with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 40 and 80 years with a confirmed diagnosis of idiopathic pulmonary fibrosis
* Both men and women must be on non-childbearing potential. Additional information regarding this requirement is available at screening.
* Capability to meet certain lung function tests at screening
* Non-smokers
* No participation in another clinical study within 4 weeks of study start.

Exclusion Criteria:

* Certain medical conditions may exclude candidates from participation.
* Blood loss or donation of 400 mL or more within 2 months of study start Significant illness (other than respiratory) within 2 weeks of study start
* Past medical personal or close family history of clinically significant ECG abnormalities
* Connective tissue disorders
* Active infection or history of systemic parasitic infection
* Known hypersensitivity to the drug.
* History of immunocompromise, including a positive HIV test result.
* History of drug or alcohol abuse within 12 months of study start
* Any condition that may compromise patient safety

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
-To investigate the possibility that some IPF patients experience increased IL-13 production. Blood samples to be collected pre-dose and weekly after dosing. -To investigate the hypothesis that QAX576 will neutralize IL-13 in patients with IPF | Week 1,2,3 and 4

SECONDARY OUTCOMES:
-To evaluate the changes in biomarkers in blood over time in patients with IPF. Serum samples will be obtained at pre-dose and 2 weeks post-dose. | Week 3

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Principal Investigator — Investigative site
Locations (6):
- United States (6):
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Clinical Trial Results for CQAX576A2202 at Novartis Clinical Trials.com — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3024